CLINICAL TRIAL: NCT05440214
Title: Targeting Emotion Dysregulation to Reduce Suicide in People With Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Peter Phalen, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1K23MH125024-01A1 (NIH)
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Psychosis; Suicide
MeSH Terms: conditions — Psychotic Disorders; Suicide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dialectical Behavior Therapy - Skill Training (Experimental)
  Interventions: Behavioral: Dialectical Behavior Therapy Skills Training
- Treatment As Usual (No Intervention)

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy Skills Training — Dialectical Behavior Therapy Skills Training (DBT-ST) is a group-based intervention focused on teaching skills for improving emotion regulation. The sessions will be offered in-person or via approved telehealth services.
  Other Names: DBT; DBT-ST; DBT Skills Group; Dialectical Behavior Therapy Skills Group
  Arms: Dialectical Behavior Therapy - Skill Training

SUMMARY:
People with psychotic disorders are excluded from most suicide-focused clinical trials despite incredibly high rates of completed suicide, and interventions that have been tested for this population have shown limited impact on suicide. Emotion dysregulation is a significant suicidogenic factor that is understudied in people with psychotic disorders. The investigators propose to implement and evaluate an intervention targeting emotion dysregulation in people with psychotic disorders while employing rigorous statistical modeling and measurement techniques including Ecological Momentary Assessment, which will support future advanced research on suicide and suicide prevention for this high-risk group.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Psychosis spectrum disorder as assessed by the Mini International Neuropsychiatric Interview (MINI) for Psychotic Disorder Studies
* Heightened suicide risk as determined by a score of 8+ on the Suicide Behaviors Questionnaire-Revised (SBQ-R). This cutoff may be revised downwards (toward lower suicide risk) if recruitment appears difficult, but will not be revised upwards.
* Enrollment and engagement in outpatient mental health services with at least one mental health service in the previous month
* 6+ grade equivalent reading level as assessed by the Wide Range Achievement Test 4 (WRAT-4)

Exclusion Criteria:

* Chart diagnosis of intellectual disability (DSM5 317, 318), traumatic brain injury, or deafness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation | Four months
  Beck Scale for Suicide Ideation. Minimum score: 0. Maximum score: 42. Higher scores are worse.
Emotion Dysregulation | Four months
  Difficulties in Emotion Regulation Scale (DERS-36). Minimum score: 36. Maximum score: 180. Higher scores are worse.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No